CLINICAL TRIAL: NCT04366050
Title: A Randomized, Double-blind, Placebo-Controlled Trial to Evaluate the Efficacy of Ramipril to Prevent ICU Admission, Need for Mechanical Ventilation or Death in Persons With COVID-19
Brief Title: Ramipril for the Treatment of COVID-19
Acronym: RAMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Rohit Loomba, Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RAMIC Trial
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ramipril 2.5mg orally daily (Experimental): Total 2.5 mg Ramipril per day once a day orally for 14 days
  Intervention: Ramipril
  Interventions: Drug: Ramipril 2.5 MG Oral Capsule
- Placebo (Placebo Comparator): Placebo in the form of a capsule, taken orally for 14 days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Ramipril 2.5 MG Oral Capsule — Include description or ramipril from protocol
  Other Names: Ramipril
  Arms: Ramipril 2.5mg orally daily
Drug: Placebo oral capsule — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
In this study we propose to treat 560 patients with ramipril or placebo for 14 days. After an initial evaluation for COVID-19 status, medical history, and symptom assessment, patients will receive either 2.5 mg/day of ramipril or placebo. Patients' symptoms and study endpoints will be monitored at regular intervals. After 14 days, patients will undergo a laboratory assessment and an end-of-treatment follow-up visit at day 28. The primary endpoints of successful therapy will be improved survival, reductions in ICU admissions, and/or reductions in use of mechanical ventilator support.

DETAILED DESCRIPTION:
Ramipril has not been studied in SARS-CoV-2 infected patients. In this study we propose to treat 560 patients with ramipril or placebo for 14 days. After an initial evaluation for COVID-19 status, medical history, and symptom assessment, patients will receive either 2.5 mg/day of ramipril or placebo. Patients' symptoms and study endpoints will be monitored at regular intervals. Additional follow-up will be performed at day 28. As an exploratory objective, biomarkers of the RAAS axis will also be monitored. The primary endpoints of successful therapy will be improved survival, reductions in ICU admissions, and/or reductions in use of mechanical ventilator support. Secondary endpoints will be the proportion of patients needing continued hospitalization, time to mortality, time to ICU admission, time to discharge from hospital, proportion of patients developing hypotension and needing pressor support, and proportion of patients developing septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to provide written informed consent prior to performing study procedures
* Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test ≤ 5 days before randomization OR Clinical presentation consistent with COVID-19 infection (fever or cough or shortness of breath) with positive IgM serology
* Currently hospitalized or in an emergency department
* Peripheral capillary oxygen saturation (SpO2) ≥ 93% on room air at screening

Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19 (use of hydroxycholoroquine or compassionate use of choloroquine or azithromycin is allowed)
* Concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2 is prohibited < 24 hours prior to study drug/placebo dosing
* Requiring mechanical ventilation at screening
* Requiring ICU care at admission
* NSAID use within 12 hours of randomization or requiring continued NSAID use during this trial
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN)
* Estimated GFR < 40 mL/min
* History of serum creatinine ≥ 2 mg/dl in the previous 28 days
* Systolic BP < 100 mm hg or diastolic BP < 65 mm hg
* Hypersensitivity to ACEI
* History of angioedema
* Outpatient use of ACE inhibitor or Angiotensin II receptor blocker in the last 7 days
* History of renal artery stenosis
* Serum potassium ≥ 5.1 mEq/L
* Pregnancy or breastfeeding
* Use of aliskiren, amifostine, lithium, sacubitril within 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Loomba, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Huang DQ, Ajmera V, Tomaszewski C, LaFree A, Bettencourt R, Thompson WK, Smith DM, Malhotra A, Mehta RL, Tolia V, Yin J, Insel PA, Leachman S, Jung J, Collier S, Richards L, Woods K, Amangurbanova M, Bhatt A, Zhang X, Penciu OM, Zarich S, Retta T, Harkins MS, Teixeira JP, Chinnock B, Utay NS, Lake JE, Loomba R. Ramipril for the Treatment of COVID-19: RAMIC, a Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Adv Ther. 2023 Nov;40(11):4805-4816. doi: 10.1007/s12325-023-02618-7. Epub 2023 Aug 24. PMID 37615850
- [Derived] Ajmera V, Thompson WK, Smith DM, Malhotra A, Mehta RL, Tolia V, Yin J, Sriram K, Insel PA, Collier S, Richards L, Loomba R. RAMIC: Design of a randomized, double-blind, placebo-controlled trial to evaluate the efficacy of ramipril in patients with COVID-19. Contemp Clin Trials. 2021 Apr;103:106330. doi: 10.1016/j.cct.2021.106330. Epub 2021 Feb 22. PMID 33631357

RESULTS

PARTICIPANT FLOW:
Groups:
- Ramipril 2.5mg Orally Daily: Total 2.5 mg Ramipril per day once a day orally for 14 days
  Intervention: Ramipril
  Ramipril 2.5 MG Oral Capsule: Include description or ramipril from protocol
Period: Overall Study
Arm/Group | Ramipril 2.5mg Orally Daily | Placebo
Started | 79 | 35
Completed | 68 | 32
Not Completed | 11 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramipril 2.5mg Orally Daily | Placebo | Total
Number analyzed (Participants) | 79 | 35 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (16) | 46 (14) | 45 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 20 | 58
  Male | 41 | 15 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 5
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 44 | 23 | 67
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 22 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Composite of Mortality or Need for ICU Admission or Ventilator Use
Description: The major primary outcome to be evaluated is improving a composite outcome of mortality or need for ICU admission or ventilator use within a 14-day window.
Time Frame: 14 days
Measure: Count of Participants; unit: Participants
Arm/Group | Ramipril 2.5mg Orally Daily | Placebo
Number analyzed (Participants) | 79 | 35
Participants | 2 | 0

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Ramipril 2.5mg Orally Daily | Placebo
All-Cause Mortality (participants affected / at risk) | 1/79 | 0/35
Serious Adverse Events (participants affected / at risk) | 2/79 | 0/35
Other Adverse Events (participants affected / at risk) | 37/79 | 19/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril 2.5mg Orally Daily (N=79) | Placebo (N=35)
Cardiopulmonary Failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramipril 2.5mg Orally Daily (N=79) | Placebo (N=35)
Lightheadedness (General disorders) | 2 (2) | 6 (6)
Diarrhea/Vomiting (Gastrointestinal disorders) | 4 (4) | 3 (3)
Drenching Sweats (General disorders) | 2 (2) | 2 (2)
Head or Body Pain (General disorders) | 6 (6) | 2 (2)
Cough/Shortness of Breath/Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Loss of Smell (General disorders) | 2 (2) | 1 (1)
Elevated Lab Markers (General disorders) | 3 (3) | 1 (1)
Cardiovascular Issues (Cardiac disorders) | 5 (5) | 0 (0)
Rectal Hemorrhage (General disorders) | 0 (0) | 1 (1)
Ear Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Steroid induced Diabetes (Endocrine disorders) | 1 (1) | 0 (0)
Worsening GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0)
Throat Swelling (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Jittery (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04366050/Prot_SAP_000.pdf